CLINICAL TRIAL: NCT06350942
Title: One Trocar-assisted Retroperitoneoscopic Ureteroureterostomy for Ureteral Duplication
Status: Completed | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Collaborators: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Principal Investigator, Nguyen Thanh Quang, Pediatric Surgeon, National Children's Hospital, Vietnam
Other Study IDs: 1451_01/BVNTW-VNCSKTE
Record Dates: First submitted 2024-03-30; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-03

CONDITIONS: Ureteral Duplication
Keywords: Duplex Kidney; Ureteral Duplication; Ureteroureterostomy; Retroperitoneoscopic; Single-trocar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Complete duplicated collecting system: The presence of two pelvicalyceal systems within a single kidney, with either obstructed or ectopic ureter
  Interventions: Procedure: one trocar-assisted retroperitoneoscopic ureteroureterostomy (OTAU)

INTERVENTIONS:
Procedure: one trocar-assisted retroperitoneoscopic ureteroureterostomy (OTAU) — A 12 mm transverse incision was made just above the iliac crest, followed by careful dissection of the fascia and muscle layer to expose the Gerota's fascia. Entry into the retroperitoneal space was achieved with a 10-mm balloon trocar, allowing for pneumoretroperitoneum establishment. Using a 10-mm laparoscope equipped with a Maryland dissector, the ureters were dissected and isolated, followed by careful exteriorization of both upper and lower pole moiety ureters with a Babcock grasper. The pathological upper pole moiety ureter was transected, preserving the normal lower pole moiety ureter and shared blood supply, and closed with a Vicryl 4/0 suture. Subsequently, an end-to-side ureteroureterostomy was performed with a 6/0 Polydioxanone running suture, with antegrade insertion of a double J stent if not previously conducted. A final retroperitoneoscopic evaluation ensured proper anastomosis alignment, and the incision was closed without drainage.

SUMMARY:
Ureteral duplication, a common anomaly affecting about 0.8% of the population, presents challenges in pediatric urology due to its diverse clinical presentations and anatomical complexity. Traditional treatments like upper pole moiety (UPM) heminephrectomy can lead to loss of renal function in the remaining lower pole moiety (LPM). Ureteroureterostomy (UU) is a safer alternative, increasingly preferred regardless of renal function or reflux presence. Minimally invasive techniques like laparoscopic and robotic procedures show promise, but robotic-assisted UU is costly, while laparoscopic UU has technical challenges. A novel approach is proposed: single-trocar retroperitoneoscopic-assisted UU, combining laparoscopic visualization advantages with simplified extracorporeal suturing, offering a promising solution for managing complete ureteral duplication. The present study was designed to describe the operative technique and outcome of OTAU in 40 cases of complete ureteral duplication in children.

DETAILED DESCRIPTION:
Ureteral duplication, a common anomaly affecting about 0.8% of the population, presents challenges in pediatric urology due to its diverse clinical presentations and anatomical complexity. Traditional treatments like upper pole moiety (UPM) heminephrectomy can lead to loss of renal function in the remaining lower pole moiety (LPM). Ureteroureterostomy (UU) is a safer alternative, increasingly preferred regardless of renal function or reflux presence. Minimally invasive techniques like laparoscopic and robotic procedures show promise, but robotic-assisted UU is costly, while laparoscopic UU has technical challenges. A novel approach is proposed: single-trocar retroperitoneoscopic-assisted UU, combining laparoscopic visualization advantages with simplified extracorporeal suturing, offering a promising solution for managing complete ureteral duplication. The present study was designed to describe the operative technique and outcome of OTAU in 40 cases of complete ureteral duplication in children.

Demographic data of patients, their clinical manifestations, classification of hydronephrosis based on the guidelines established by the Society for Fetal Urology (SFU), dimensions of the renal pelvis measured in the anterior-posterior direction (APD), diameters of the ureters, duration of surgical procedures, duration of hospitalization, and subsequent follow-up information were systematically gathered prospectively to evaluate the long-term outcomes of the proposing surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ureteral duplication.
* Age no more than 18 years old
* The surgical technique performed must be one trocar-assisted retroperitoneoscopic ureteroureterostomy.
* Followed up at least 2-4 years

Exclusion Criteria:

* Patients exhibiting reflux to the ureter of the lower pole moiety (LPM)
* Patients with prior urologic surgeries or other urological anomalies

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients diagnosed with ureteral duplication, including with either ectopic or obstructed ureter, were treated with OTAU between September 2016 and December 2020. Preoperative diagnostic evaluations included blood tests, urinalysis, culture, renal ultrasonography (US), and voiding cystourethrogram to identify vesicoureteral reflux. Dimercaptosuccinic acid (DMSA) scintigraphy was used to measure the differential renal function (DRF). UU was performed irrespective of the differential function of the upper pole moiety (UPM) or the patient's age.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Mean operating time | through study completion (4 years)
  The average operating time (minutes) of OTAU
Intraoperative complications | through study completion (4 years)
  Complications experienced during the procedure
Conversion to open | through study completion (4 years)
  Incidence in which the operation must be switch to open surgery
Early postoperative complications | through study completion (4 years)
  Complications after OTAU including UTI and wound infection
Median length of hospital stays | through study completion (4 years)
  Average time (days) the patient has to stay at the hospital post-operation
Mean UPM renal pelvis' APD | through study completion (4 years)
  The average anterior-posterior diameter (mm) of the upper pole moiety before and after the operation
Mean SFU of UPM renal pelvis | through study completion (4 years)
  The average Society of Fetal Urology classification of the upper pole moiety before and after the operation
Mean UPM ureter's diameter | through study completion (4 years)
  The average ureter's diameter (mm) of the upper pole moiety before and after the operation
Mean UPM DRF | through study completion (4 years)
  The average differential renal function (%) (measurement of each kidney's ability to extract tracer from blood) of the upper pole moiety before and after operation
Mean DRF of operated side | through study completion (4 years)
  The average differential renal function (%) of the operated side before and after operation

CONTACTS AND LOCATIONS:
Overall Officials: Quang T Nguyen, M.D., Principal Investigator — : Department of Pediatric Surgery, The National Hospital of Pediatrics, Hanoi, Vietnam
Locations (2):
- Vietnam (2):
  - The National Hospital of Pediatrics, Hanoi
  - Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glassberg KI, Braren V, Duckett JW, Jacobs EC, King LR, Lebowitz RL, Perlmutter AD, Stephens FD. Suggested terminology for duplex systems, ectopic ureters and ureteroceles. J Urol. 1984 Dec;132(6):1153-4. doi: 10.1016/s0022-5347(17)50072-5. PMID 6502807
- [Background] Chacko JK, Koyle MA, Mingin GC, Furness PD 3rd. Ipsilateral ureteroureterostomy in the surgical management of the severely dilated ureter in ureteral duplication. J Urol. 2007 Oct;178(4 Pt 2):1689-92. doi: 10.1016/j.juro.2007.05.098. Epub 2007 Aug 17. PMID 17707022
- [Background] Fernbach SK, Feinstein KA, Spencer K, Lindstrom CA. Ureteral duplication and its complications. Radiographics. 1997 Jan-Feb;17(1):109-27. doi: 10.1148/radiographics.17.1.9017803.
- [Background] Stokland E, Jodal U, Sixt R, Swerkersson S, Hansson S. Uncomplicated duplex kidney and DMSA scintigraphy in children with urinary tract infection. Pediatr Radiol. 2007 Aug;37(8):826-8. doi: 10.1007/s00247-007-0518-x. Epub 2007 Jun 26. PMID 17593362
- [Background] Timberlake MD, Corbett ST. Minimally invasive techniques for management of the ureterocele and ectopic ureter: upper tract versus lower tract approach. Urol Clin North Am. 2015 Feb;42(1):61-76. doi: 10.1016/j.ucl.2014.09.006. Epub 2014 Oct 11. PMID 25455173
- [Background] McLeod DJ, Alpert SA, Ural Z, Jayanthi VR. Ureteroureterostomy irrespective of ureteral size or upper pole function: a single center experience. J Pediatr Urol. 2014 Aug;10(4):616-9. doi: 10.1016/j.jpurol.2014.05.003. Epub 2014 Jun 2. PMID 24947344
- [Background] Lashley DB, McAleer IM, Kaplan GW. Ipsilateral ureteroureterostomy for the treatment of vesicoureteral reflux or obstruction associated with complete ureteral duplication. J Urol. 2001 Feb;165(2):552-4. doi: 10.1097/00005392-200102000-00067. PMID 11176433
- [Background] Prieto J, Ziada A, Baker L, Snodgrass W. Ureteroureterostomy via inguinal incision for ectopic ureters and ureteroceles without ipsilateral lower pole reflux. J Urol. 2009 Apr;181(4):1844-8; discussion 1848-50. doi: 10.1016/j.juro.2008.12.004. Epub 2009 Feb 23. PMID 19233406
- [Background] Cundy TP, Shetty K, Clark J, Chang TP, Sriskandarajah K, Gattas NE, Najmaldin A, Yang GZ, Darzi A. The first decade of robotic surgery in children. J Pediatr Surg. 2013 Apr;48(4):858-65. doi: 10.1016/j.jpedsurg.2013.01.031. PMID 23583146
- [Background] Herz D, Smith J, McLeod D, Schober M, Preece J, Merguerian P. Robot-assisted laparoscopic management of duplex renal anomaly: Comparison of surgical outcomes to traditional pure laparoscopic and open surgery. J Pediatr Urol. 2016 Feb;12(1):44.e1-7. doi: 10.1016/j.jpurol.2015.04.046. Epub 2015 Aug 17. PMID 26443241
- [Background] Wong NC, Braga LH. Open ureteroureterostomy for repair of upper-pole ectopic ureters in children with duplex systems: is stenting really necessary? J Pediatr Urol. 2019 Feb;15(1):72.e1-72.e7. doi: 10.1016/j.jpurol.2018.10.014. Epub 2018 Oct 24. PMID 30477994
- [Result] Gonzalez R, Piaggio L. Initial experience with laparoscopic ipsilateral ureteroureterostomy in infants and children for duplication anomalies of the urinary tract. J Urol. 2007 Jun;177(6):2315-8. doi: 10.1016/j.juro.2007.01.177. PMID 17509348
- [Result] Lowe GJ, Canon SJ, Jayanthi VR. Laparoscopic reconstructive options for obstruction in children with duplex renal anomalies. BJU Int. 2008 Jan;101(2):227-30. doi: 10.1111/j.1464-410X.2007.07106.x. Epub 2007 Sep 13. PMID 17868427
- [Result] Chandrasekharam V, Jayaram H. Laparoscopic ipsilateral ureteroureterostomy for the management of children with duplication anomalies. J Indian Assoc Pediatr Surg. 2015 Jan;20(1):27-31. doi: 10.4103/0971-9261.145442. PMID 25552828
- [Result] Storm DW, Modi A, Jayanthi VR. Laparoscopic ipsilateral ureteroureterostomy in the management of ureteral ectopia in infants and children. J Pediatr Urol. 2011 Oct;7(5):529-33. doi: 10.1016/j.jpurol.2010.08.004. Epub 2010 Sep 25. PMID 20869918
- [Result] Lee NG, Corbett ST, Cobb K, Bailey GC, Burns AS, Peters CA. Bi-Institutional Comparison of Robot-Assisted Laparoscopic Versus Open Ureteroureterostomy in the Pediatric Population. J Endourol. 2015 Nov;29(11):1237-41. doi: 10.1089/end.2015.0223. Epub 2015 Aug 21. PMID 26159231
- [Result] Kawal T, Srinivasan AK, Talwar R, Chu DI, Long C, Weiss D, Van Batavia J, Kolon TF, Shukla AR. Ipsilateral ureteroureterostomy: does function of the obstructed moiety matter? J Pediatr Urol. 2019 Feb;15(1):50.e1-50.e6. doi: 10.1016/j.jpurol.2018.08.012. Epub 2018 Aug 20. PMID 30243559
- [Result] Biles MJ, Finkelstein JB, Silva MV, Lambert SM, Casale P. Innovation in Robotics and Pediatric Urology: Robotic Ureteroureterostomy for Duplex Systems with Ureteral Ectopia. J Endourol. 2016 Oct;30(10):1041-1048. doi: 10.1089/end.2015.0645. Epub 2016 Sep 16. PMID 27542552
- [Result] Liem NT, Dung LA, Viet ND. Single trocar retroperitoneoscopic assisted ipsilateral ureteroureterostomy for ureteral duplication. Pediatr Surg Int. 2012 Oct;28(10):1031-4. doi: 10.1007/s00383-012-3158-7. Epub 2012 Aug 12. PMID 22885733
- [Result] Grimsby GM, Merchant Z, Jacobs MA, Gargollo PC. Laparoscopic-assisted ureteroureterostomy for duplication anomalies in children. J Endourol. 2014 Oct;28(10):1173-7. doi: 10.1089/end.2014.0113. Epub 2014 Aug 13. PMID 25010444
- [Result] Bieri M, Smith CK, Smith AY, Borden TA. Ipsilateral ureteroureterostomy for single ureteral reflux or obstruction in a duplicate system. J Urol. 1998 Mar;159(3):1016-8. PMID 9474221